CLINICAL TRIAL: NCT06717789
Title: Post-Market Prospective Clinical Follow Up Study on the Symptomatic Treatment of Musculoskeletal Pain Through Sensory Nerve Stimulation Using the Compex SP8.0 Device
Brief Title: Compex SP8.0 - Symptomatic Treatment of Musculoskeletal Pain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: DJO UK Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ENOVIS-S-INP-0006
Record Dates: First submitted 2024-11-29; First posted 2024-12-05 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2024-11

CONDITIONS: Musculoskeletal Conditions; Musculoskeletal Pain
Keywords: Electrostimulation; Transcutaneous Electrical Nerve Stimulation (TENS); Stimulation of sensory nerves; Compex SP8.0; Gate control principle; Endorphinic TENS; Low Frequency TENS; High Frequency TENS
MeSH Terms: conditions — Musculoskeletal Pain | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Intervention Model Description: Transcutaneous Electrical Nerve Stimulation (TENS) with the Compex SP8.0 device
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Frequency TENS (Experimental): Based on the diagnosis and the type of pain , subjects will be assigned to the High Frequency TENS (gate control principle at 50-150 Hz) treatmet group, which includes the following preset programs:
  * Pain management TENS
  * Epicondylitis
  * Tendinitis.
  Interventions: Device: Transcutaneous Electrical Nerve Stimulation (TENS) with the Compex SP8.0 device
- Low frequency TENS (Experimental): Based on the diagnosis and the type of pain , subjects will be assigned to the Low Frequency TENS (endorphinic TENS at 5 Hz) treatmet group, which includes the following preset programs:
  * Muscle pain
  * Neck pain
  * Back pain
  Interventions: Device: Transcutaneous Electrical Nerve Stimulation (TENS) with the Compex SP8.0 device

INTERVENTIONS:
Device: Transcutaneous Electrical Nerve Stimulation (TENS) with the Compex SP8.0 device — Transcutaneous Electrical Nerve Stimulation (TENS) with the Compex SP8.0 device, using the following pain management program,
  • High Intensity TENS (50-150 Hz)
  Arms: High Frequency TENS
Device: Transcutaneous Electrical Nerve Stimulation (TENS) with the Compex SP8.0 device — Transcutaneous Electrical Nerve Stimulation (TENS) with the Compex SP8.0 device, using the following pain management program,
  • Low Intensity TENS (5 Hz)
  Arms: Low frequency TENS

SUMMARY:
This post-market clinical study of the SP8.0 Compex device aims to comprehensively assess the safety and performance of the device when used in accordance with the approved Instructions for Use. The results of this study will also support the clinical evaluation of the next-generation wireless product currently under development.

The Compex Consumer devices contain different programs, such as conditioning, fitness, recovery, massage, rehabilitation, and pain management.

This study will utilize the Compex SP 8.0 pain management programs, with the aim of assessing the effectiveness of the treatment provided by the device in managing pain through different physiological mechanisms.

DETAILED DESCRIPTION:
Subjects will be treated with the Compex device according to the intended use of the device and as per routine clinical practice. Clinical data will be collected in healthcare settings as part of the routine clinical practice and according to the study protocol. Additional data points will be recorded pre and post use of the advised treatment with the compex device using an electronic patient diary.

Adult subjects who require symptomatic treatment of musculoskeletal pain (nociceptive pain or neuropathic/nociplastic pain), with a Numeric Pain Rating Scale (NPRS) score of 4 or more at baseline will undergo Electrical Nerve Stimulation with the Compex SP8.0 device at home for up to 4 weeks.

The investigator will train subjects on how to use the device at home and a guide will be provided to each subject to help them when using the device at home.

For all subjects the first treatment session will be performed by the investigator at the clinic.

The assessment of pain level will be completed by the investigator during onsite visits: before treatment (Baseline Visit), after 2 weeks of treatment and at the 4 weeks/End of study visit. Additionally, subjects will be asked to record their level of pain before and immediately after each treatment session on an electronic diary.

The assessment of the pain level experienced by the subjects will be performed using the Numeric Pain Rating Scale (NPRS). Subjects will be asked to rate the level of pain using a 0-10 scale, with zero meaning "no pain" and 10 meaning "the worst pain imaginable".

The tests used to assess symptoms, compliance with treatment and satisfaction/usability of the device are:

1. Numeric Pain Rating Scale (NPRS) on a 0 to 10 scale
2. Usability/Satisfaction Questionnaire on a 4-point Likert scale
3. Electronic Compliance diary

Participants will be stratified based on their type of pain (nociceptive vs. neuropathic/nociplastic) and then assigned within strata to one of the treatment groups: TENS HIGH FREQUENCY (50-150Hz) or TENS LOW FREQUENCY (5Hz) The diagnosis of the type of pain experienced by individual subjects will be performed by the investigator based on symptoms and physical examination in routine practice.

Subjects suffering from chronic musculoskeletal pain will be allocated to the low frequency TENS group, those with acute neurogenic pain will be allocated to the high frequency TENS group.

The following programs of pain management will be used according to the subjects assigned group:

PROGRAMMING BASIC FREQUENCY TOTAL TIME PAIN MANAGEMENT TENS 50-150Hz 20 min EPICONDYLITIS/TENDINITIS 50-150Hz 20 min MUSCLE/NECK/BACK PAIN 5Hz 20 min

The treatment with the Compex SP8.0 devices can be performed in addition to subjects prescribed rehabilitation exercises and during their functional activities.

The recommendation would be to have 2 treatment sessions per day for a total of 4 weeks or until full recovery (Pain scored 0 on the NPRS). The minimum number of accepted treatments is at least 6 treatments per week. A lower number of sessions per week (less than 6 per week) will prompt the subjects to be considered in the intention to treat population but not in the per protocol data set.

Subjects will be instructed to use the mi-function for each treatment session to optimize the treatment settings.

Subjects will be asked to record each treatment session performed and pain scores experienced before and after treatment, on the subject's diary, in order to assess daily compliance to the scheduled treatment plan and to evaluate the instant and short-term effect of the treatment.

The subjects will be evaluated at the study site for 4 scheduled onsite visits and 2 phone contacts as detailed in the study flowchart.

Follow-up phone calls with the subjects will be performed on a regular basis. During the 4 weeks of treatment, 1 phone call per week will be performed with exception of the weeks when an onsite visit is scheduled. These regular contacts serve to remind the subject to follow the treatment plan and to complete the compliance diary. Additionally, during each phone call check-in, subjects will be asked to report if any issues/adverse events have occurred since the last visit or phone contact. The regular phone contact with subjects should help in keeping the adherence to the protocol and have a higher compliance to the treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Adult subjects currently experiencing musculoskeletal pain with a Numeric Pain Rating Scale (NPRS) score of 4 or more at baseline.
2. Subjects are considered suitable to self-administer stimulation of motor nerves or stimulation of sensory nerves at home, based on the Investigator's judgement.
3. Subjects are suitable to receive treatment using the Compex SP8.0 device Pain management programs (pre-set parameters) for up to 4 weeks, based on the Investigator's judgement.
4. Subject, both male and female, ≥ 18 years of age at the time of consent
5. Subject has reviewed the IEC-approved consent form, has properly consented per the protocol and has documented their consent to participate in the study by signing the Ethics-approved consent form.
6. Subject does not meet any of the exclusion criteria

Exclusion Criteria:

1. Pregnancy
2. Presence of Implanted electronic devices (e.g., pacemakers, defibrillators)
3. Skin conditions that contraindicate TENS use (e.g., rashes, wounds in electrode placement areas).
4. Known allergy to electrode materials.
5. Current participation in another clinical study that could interfere with this study's outcomes.
6. Subjects who are not able to read and understand the Instructions for Use, warnings, cautions and dangers
7. Subjects who are not able to read and understand indications and contraindications of the device
8. Subjects who are not able to sense auditory and visual signals
9. Subjects who are being treated with any other electrotherapy device for pain relief.
10. Subjects who are being treated with acupuncture
11. Participation in another clinical study within 30 days prior to screening

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Change in pain level | From enrollment to full recovery or end of treatment at week 4
  Improvement in pain demonstrated by the score on the Numerical Pain Rating Scale (NPRS) at the beginning and the end of the treatment period when using the pain management treatment programs of the device.
  The Numerical Pain Rating scale (NRS)is a 0-10 scale, with zero meaning "no pain" and 10 meaning "the worst pain imaginable".
  The overall success of the study as well as the evaluation of the primary endpoint will be based on the proportion of subjects who experience a ≥ 2-point decrease in pain scores at the end of the treatment period as compared to baseline.

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | From enrollment to full recovery or end of treatment at week 4
  Adverse events/malfunctions/complications reported during the study. Subjects and Investigators will be prompted to record such issues on the AE evaluation form. The incidence of the observed events will be tabulated by category (as in No. of observed events / No. of patients in the safety population).

OTHER OUTCOMES:
Device Usability and subject's satisfaction | From enrollment to full recovery or end of treatment at week 4
  Evaluation of device usability by the subjects and subjects' satisfaction on a 4-point Likert Scale. Subjects can choose the option that best corresponds with how they feel about the question,
Short term effects of the treatment on pain level | From enrollment to full recovery or end of treatment at week 4
  Evaluation of the immediate improvement of pain using the NPRS following each daily treatment.
  The Numerical Pain Rating scale (NRS)is a 0-10 scale, with zero meaning "no pain" and 10 meaning "the worst pain imaginable".
  The efficacy data for this analysis will consist of data obtained from the patient diaries.

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Pigott, Principal Investigator — Salford University Sports Injury Clinic
Locations (2):
- United Kingdom (2):
  - Salford University Sports Injury Clinic, Salford, Manchester
  - Worsley Physiotherapy and Sports Injuries Clinic, Worsley, Manchester

IPD SHARING:
Plan to Share IPD: No